CLINICAL TRIAL: NCT01085162
Title: An Open-Label Prospective, Non-Randomized, International, Multi-center, Long-term Follow-up Study to Evaluate the Predictive Value of BMS747158 Positron Emission Tomography (PET) Myocardial Perfusion Imaging (MPI) in Patients Suspected of Coronary Artery Disease (CAD)
Brief Title: A Long-term Follow-up Study to Evaluate the Predictive Value of BMS747158 in Patients Suspected of Coronary Artery Disease (CAD)
Status: Withdrawn | Type: Observational
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: BMS747158-501
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary Artery Disease; PET imaging; SPECT imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — BMS 747158-02

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BMS747158 — BMS747158 is a novel PET MPI agent labeled with Fluorine-18.

SUMMARY:
This long-term study will follow patients with known or suspected of having coronary artery disease (CAD) and have participated in present and future BMS747158 clinical studies. The purpose of this study is to evaluate the long-term predictive value associated with BMS747158 Positron Emission Tomography (PET) Myocardial Perfusion Imaging (MPI).

ELIGIBILITY:
Inclusion Criteria:

* Have known or suspected CAD
* Have participated in a BMS747158 clinical study
* Have received at least 1 dose of BMS747158
* Provide signed informed consent for this study prior to any follow-up contact
* Be capable of communicating effectively with study personnel

Exclusion Criteria:

* If determined by the Investigator that participation in the study is not in the best interest of the patient or for any sound medical, psychiatric, and/or social reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from prior BMS747158 clinical studies. They will have known or suspected CAD and have received at least 1 dose of BMS747158.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Independent predictive value of BMS747158 PET MPI | 2 years
  The primary outcome measure is the independent predictive value (PV) of rest and stress BMS747158 PET MPI in defining cardicac populations at high and low risk of developing cardiac events.

SECONDARY OUTCOMES:
Comparison of independent incremental PV of BMS747158 PET MPI to SPECT MPI | 2 years
  Comparison of independent incremental PV of BMS747158 PET MPI to that of single photon SPECT MPI in patients with known or suspected CAD
Incidence of soft and hard cardiac events post BMS747158 administration | 2 years
  Incidence of soft and hard cardiac events post BMS747158 administration in patients with positive and negative BMS747158 PET MPI scans obtained in the qualifying study

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, S. Mark Taper Foundation Imaging Center, Los Angeles, California, United States

REFERENCES:
- [Background] Clark AN, Beller GA. The present role of nuclear cardiology in clinical practice. Q J Nucl Med Mol Imaging. 2005 Mar;49(1):43-58. PMID 15724135
- [Background] Ritchie JL, Bateman TM, Bonow RO, Crawford MH, Gibbons RJ, Hall RJ, O'Rourke RA, Parisi AF, Verani MS. Guidelines for clinical use of cardiac radionuclide imaging: A report of the American College of Cardiology/American Heart Association Task Force on assessment of diagnostic and therapeutic cardiovascular procedures (Committee on Radionuclide Imaging)--developed in collaboration with the American Society of Nuclear Cardiology. J Nucl Cardiol. 1995 Mar-Apr;2(2 Pt 1):172-92. doi: 10.1016/s1071-3581(06)80030-9. No abstract available. PMID 9463028
- [Background] Di Carli MF, Hachamovitch R. New technology for noninvasive evaluation of coronary artery disease. Circulation. 2007 Mar 20;115(11):1464-80. doi: 10.1161/CIRCULATIONAHA.106.629808. No abstract available. PMID 17372188
- [Background] Glover DK, Gropler RJ. Journey to find the ideal PET flow tracer for clinical use: are we there yet? J Nucl Cardiol. 2007 Nov-Dec;14(6):765-8. doi: 10.1016/j.nuclcard.2007.09.019. No abstract available. PMID 18022101
- [Background] Beller GA, Zaret BL. Contributions of nuclear cardiology to diagnosis and prognosis of patients with coronary artery disease. Circulation. 2000 Mar 28;101(12):1465-78. doi: 10.1161/01.cir.101.12.1465. No abstract available. PMID 10736294
- [Background] Beller GA. First annual Mario S. Verani, MD, Memorial lecture: clinical value of myocardial perfusion imaging in coronary artery disease. J Nucl Cardiol. 2003 Sep-Oct;10(5):529-42. doi: 10.1016/s1071-3581(03)00655-x. PMID 14569247
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):e21-181. doi: 10.1161/CIRCULATIONAHA.108.191261. Epub 2008 Dec 15. No abstract available. PMID 19075105